CLINICAL TRIAL: NCT05257174
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Jing Si Herbal Tea Liquid Packets on Fatigue in Patients With Inflammatory Arthritis
Brief Title: The Effects of Jing Si Herbal Tea Liquid Packets on Fatigue in Patients With Inflammatory Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB110-301-A
Record Dates: First submitted 2022-01-28; First posted 2022-02-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Arthritis; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Fatigue
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jing Si Herbal Tea LIQUID PACKETS (Experimental): one packet oral twice daily for three months
  Interventions: Dietary Supplement: Jing Si Herbal Tea LIQUID PACKETS
- Placebo (Placebo Comparator): one packet oral twice daily for three months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Jing Si Herbal Tea LIQUID PACKETS — intake Jing Si Herbal Tea LIQUID PACKETS twice daily for three months
  Arms: Jing Si Herbal Tea LIQUID PACKETS
Dietary Supplement: Placebo — intake Placebo twice daily for three months
  Arms: Placebo

SUMMARY:
Fatigue is a common feature in patients with rheumatic conditions. Fatigue can lead to a decline in physical function, self-confidence, cognitive status, and work performance and significantly impact the quality of life. While pain and inflammation of arthritis can be well controlled nowadays attributed to the advances in anti-rheumatic medications, fatigue remains a challenge. Even with proper therapies for arthritis, the prevalence of severe fatigue is more than 30%, which is a significant burden to both physicians and patients. However, there is no regimen to alleviate fatigue among patients with inflammatory arthritis. Finding a way to combat fatigue will significantly help improve patients' physical and mental state and family society.

To investigate the efficacy of Jing Si Herbal Tea Liquid Packets on fatigue in patients with inflammatory arthritis, the investigators propose a two-year research project to recruit approximately 150 patients with fatigue and inflammatory arthritis, including rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis. This project is designed as a randomized, double-blind, placebo-controlled study. The recruited patients will be randomized to receive Jing Si Herbal Tea Liquid Packets or a matching placebo in combination with the background regular anti-rheumatic therapy. The severity of fatigue will be obtained by questionnaire. Clinical parameters, including demographic data and disease activities, will be collected during each visit.

ELIGIBILITY:
Inclusion Criteria:

* inflammatory arthritis, any of the following diagnosis

  1. Rheumatoid arthritis, based on ACR (American College of Rheumatology) classification criteria
  2. Ankylosing spondylitis, based on modified New York Criteria
  3. Psoriatic arthritis, based on 2006 CASPAR (ClASsification criteria for Psoriatic ARthritis) criteria

Exclusion Criteria:

1. active infection or chronic infection
2. uncontrolled disease status of inflammatory arthritis
3. unwilling to take herbal tea
4. with difficulty for return visits

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in level of fatigue [Time Frame: 4, 8, 12 weeks after Jing Si Herbal Tea Liquid Packets] | Change of fatigue level every 4 weeks until 12 weeks after Jing Si Herbal Tea Liquid Packets
  Fatigue assessment measured by the functional assessment of chronic illness Therapy- Fatigue (FACIT- F) (0-52; higher score=less fatigue)

SECONDARY OUTCOMES:
Change in disease activity of inflammatory arthritis [Time Frame: 4, 8, 12 weeks after Jing Si Herbal Tea Liquid Packets] | Change of disease activity every 4 weeks until 12 weeks after Jing Si Herbal Tea Liquid Packets
  Disease activity of inflammatory arthritis measured by the Disease Activity Score based on 28 joints (DAS28) (0-9.55; higher score=more active) for rheumatoid arthritis, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (0-10; higher score=more active) for ankylosing spondylitis, and Disease Activity in PSoriatic Arthritis (DAPSA) (0-204; higher score=more active) for psoriatic arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Ying Su, MD,PhD, Principal Investigator — Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in fatigue among patients with inflammatory arthritis. Data or samples shared will be coded, with no PHI (protected health information) included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.

REFERENCES:
- [Background] Overman CL, Kool MB, Da Silva JA, Geenen R. The prevalence of severe fatigue in rheumatic diseases: an international study. Clin Rheumatol. 2016 Feb;35(2):409-15. doi: 10.1007/s10067-015-3035-6. Epub 2015 Aug 15. PMID 26272057
- [Background] Esbensen BA, Stallknecht SE, Madsen ME, Hagelund L, Pilgaard T. Correlations of fatigue in Danish patients with rheumatoid arthritis, psoriatic arthritis and spondyloarthritis. PLoS One. 2020 Aug 3;15(8):e0237117. doi: 10.1371/journal.pone.0237117. eCollection 2020. PMID 32745130